CLINICAL TRIAL: NCT04605783
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate A Dietary Supplement to Maintain Gut Health During Deployment and Travel
Brief Title: Trial to Evaluate Dietary Supplements to Maintain Gut Health During Travel
Acronym: P2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IDCRP-123
Record Dates: First submitted 2020-09-16; First posted 2020-10-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diarrhea
Keywords: Diarrhea, Prevention, Deployment, Supplements
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized, placebo-controlled, double-blind clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Travelan® (Experimental): Product will be started 2 days prior to arrival in overseas destination and maintained for a maximum duration of 20 days (minimum of 10 days) during travel or deployment.
  Interventions: Dietary Supplement: Travelan®
- Placebo (Placebo Comparator): Placebo will be started 2 days prior to arrival in overseas destination and maintained for a maximum duration of 20 days (minimum of 10 days) during travel or deployment.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Travelan® — Travelan® (600mg) taken as 1 sachet twice daily with meals. Product will be started 2 days prior to arrival and maintained for a maximum duration of 20 days (minimum of 10 days) during travel or deployment.
  Arms: Travelan®
Other: Placebo — Maltodextrin - To be started 2 days prior to arrival and maintained for a maximum duration of 20 days (minimum of 10 days) during travel or deployment.
  Arms: Placebo

SUMMARY:
Passive immunoprophylaxis is a class of dietary supplements that is lawfully marketed in the US for maintenance of gut health (GH). This randomized, double-blind, clinical trial will evaluate passive immunoprophylaxis (Travelan®) product compared with placebo, to assess the ability to maintain normal gut function during travel. The results of this clinical trial will be used to evaluate the use of a dietary supplement to maintain GH during deployment and travel and is not intended to support a marketing application of any dietary supplement as a drug or biological product for human use.

DETAILED DESCRIPTION:
Probiotics and passive immunoprophylaxis are classes of dietary supplements that are lawfully marketed in the US for maintenance of gut health (GH). This randomized, double-blind, clinical trial will evaluate one commercially available dietary supplement products (passive immunoprophylaxis (Travelan®), compared with placebo, to assess their ability to maintain normal gut function during travel. The results of this clinical trial will be used to evaluate the use of Travelan® to maintain GH during deployment and travel and is not intended to support a marketing application of any dietary supplement as a drug or biological product for human use. This study is a multi-site, randomized, placebo-controlled, double-blind clinical trial conducted on travelers and deployed US and United Kingdom (UK) military personnel. The study will test Travelan®, compared with placebo for maintenance of GH during and immediately after travel. Enrollment of 868 deployed military personnel or travelers will occur at sites within the Uniformed Services University of the Health Sciences (USU) Infectious Disease Clinical Research Program (IDCRP) network and the UK military. Subjects will be randomized to receive a masked regimen of Travelan® or placebo taken as 1 sachet twice daily with meals. Chemoprophylaxis will be started 2 days prior to arrival and maintained for a maximum duration of 20 days (minimum of 10 days) during travel or deployment. Stool smears collected during travel will be used for evaluating the microbiome and for gut pathogen identification. Paired (pre and post-supplement administration) sera and stool samples (pre- and post-supplement administration) will be collected for testing of exploratory objectives. Primary Endpoint (Efficacy): The primary efficacy endpoint is the combined endpoint of incidence of GH disruption (defined as 3 or more unformed stools in a 24-hour period) OR 2 or more unformed stools and one or more associated symptoms (nausea, vomiting, abdominal pain, fever, bloody stool) in a 24-hour period OR antibiotic treatment for diarrhea per subject report, during the period of prophylaxis. Primary endpoint data will be obtained from review of the Travel Diary. Secondary Objectives: Secondary endpoints will include an evaluation of compliance with each dietary supplement and tolerability (e.g. taste, bloating, flatulence, etc.); these will be assessed using the Travel Diary. Differences in GH associated enteropathogen distribution among the 2 treatment groups will be determined by testing stool smears collected by subjects during a GH deficit using a polymerase chain reaction (PCR) assay. Exploratory objectives related to changes in the gut microbiome with dietary supplement use and proteomic signatures of the host-pathogen interaction will be addressed contingent on the availability of additional funding.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old, able to read and speak English fluently and provide informed consent
* Travel or deployment with minimum of 10 consecutive days at intermediate to high risk for GH disruption destination (not counting quarantine period)
* Ability to complete a follow-up visit following return from travel
* Ability to provide a stool sample prior to start of prophylaxis
* Willingness to comply with study procedures

Exclusion Criteria:

* Subject-reported history of any known functional bowel disorder (including Irritable Bowel Syndrome) or chronic gastrointestinal disease (e.g. Inflammatory Bowel Disease) which in the opinion of the investigator would preclude assessment of study outcomes
* Antibiotic use within 7 days prior to start of prophylaxis (except for malaria prophylaxis including doxycycline, chloroquine, atovaquone/proguanil, mefloquine, primaquine, and tafenoquine)
* Experiencing diarrheal illness (defined as 3 or more loose/liquid stools in a 24 hour period) within 3 days prior to start of prophylaxis
* Planned use of any investigational or non-registered drug, antibiotic or other probiotics or prebiotics (outside of the study product) during the study period. This does not include consumption of yogurt products
* Intended use of a GH disruption prophylactic (e.g. Pepto-Bismol, rifaximin) during the study period
* Any planned medication usage during the study period that is deemed by the PI to interfere with GI function including but not limited to anti-diarrheals and prokinetics
* Any confirmed or suspected cancer, or use of immunosuppressant medication (topical steroids are permitted) in the last 6 months which in the opinion of the investigator would impair interpretation of the study data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of gut health deficiencies | up to 20 days
  Combined endpoint of incidence of GH deficiencies (defined as 3 or more unformed stools in a 24-hour period) OR 2 or more unformed stools and one or more associated symptoms (nausea, vomiting, abdominal pain, fever, bloody stool) in a 24-hour period OR antibiotic treatment for diarrhea per subject report, during the period of prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: David R Tribble, MD, DrPH, Principal Investigator — Infectious Disease Clinical Research Program, Uniformed Services University of the Health Sciences
Locations (6):
- United States (4):
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Naval Medical Center Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
- United Kingdom (2):
  - United Kingdom Ministry of Defence, Birmingham
  - The Liverpool School of Tropical Medicine- Well Travelled Clinic, Liverpool

IPD SHARING:
Plan to Share IPD: No